CLINICAL TRIAL: NCT02491554
Title: Deep braIn Stimulation for Tremor TractographIC Versus Traditional
Acronym: DISTINCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Medtronic Neuromodulation Europe (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Volker Arnd Coenen, Prof. Dr. med., University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P000847; DRKS00008913 (Registry Identifier: German Clinical Trial Register)
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Essential Tremor
Keywords: Deep Brain Stimulation; Essential tremor; DISTINCT; MR-tractography guided DBS implantation; Conventional AC-PC based DBS implantation
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional AC-PC based implantation of ACTIVA INS DBS system (Active Comparator): Conventional AC-PC based DBS implantation in the thalamic/subthalamic region (Vim-cZI) starting as awake surgery with a brief general anesthesia for stimulator implantation at the end of surgery.
  Interventions: Device: Conventional AC-PC based implantation of ACTIVA INS DBS system
- MR-tractography guided implantation of ACTIVA INS DBS system (Experimental): MR-tractography guided DBS implantation in the dentato-rubro-thalamic bundle (DRT) in general anesthesia.
  Interventions: Device: MR-tractography guided implantation of ACTIVA INS DBS system

INTERVENTIONS:
Device: Conventional AC-PC based implantation of ACTIVA INS DBS system — Conventional AC-PC based implantation of ACTIVA INS DBS system (manufactured by Medtronic) in the thalamic/subthalamic region (Vim-cZI).
  Other Names: Medtronic ACTIVA INS Deep Brain Stimulation system
  Arms: Conventional AC-PC based implantation of ACTIVA INS DBS system
Device: MR-tractography guided implantation of ACTIVA INS DBS system — MR-tractography guided implantation of ACTIVA INS DBS system (manufactured by Medtronic) in the DRT.
  Other Names: Medtronic ACTIVA INS Deep Brain Stimulation system
  Arms: MR-tractography guided implantation of ACTIVA INS DBS system

SUMMARY:
This is a monocentric, randomized, controlled, 2 arms, interventional, observer-blinded feasibility trial.

Patients suffering from essential tremor (ET) will be treated with Deep Brain Stimulation (DBS). For the implantation of the DBS electrodes and the DBS system (Activa INS, Medtronic) patients will randomized either to conventional stereotactic surgery of thalamic/subthalamic region with short anesthesia or to MR-tractography guided stereotactic surgery with target point of the dentato-rubro-thalamic bundle (DRT) in general anesthesia.

Patients will visit the study center at screening, baseline/neurosurgery, six and twelve months after neurosurgery.

DETAILED DESCRIPTION:
In this monocentric, randomized, controlled, 2 arms, interventional, observer-blinded feasibility trial patients suffering from therapy resistant essential tremor (ET) will be treated with Deep Brain Stimulation (DBS).

After screening (e.g. obtaining informed consent, assessment of inclusion/exclusion criteria etc.) patients will be randomized to one of the following groups:

Group 1 (conventional):

Conventional AC-PC based DBS implantation in the thalamic/subthalamic region (Vim-cZI) starting as awake surgery with a brief general anesthesia for stimulator implantation at the end of surgery.

Group 2 (tractographic):

Magnetic resonance (MR)-tractography guided DBS implantation in the dentato-rubro-thalamic bundle (DRT) in general anesthesia

At the baseline/neurosurgery visit Quality of Life (QoL) and other parameters will assessed. Medtronic's Activa INS DBS will be implanted according to randomization. DBS will be started approximately one month after surgery and will be applied as per routine.

Patients will have their routine visits. For this trial data of the (routine) visits six and twelve months after neurosurgery will be collected.

Patients receive DBS after the end of the trial according to local standards.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 25 and ≤ 80 years
2. Patients with Essential Tremor according to the criteria of the consensus statement of the movement disorders society (Deuschl et al. 1998) are included with a medical treatment resistant and disabling postural and/or intentional tremor.
3. FTMTRS to be completed within 42 days prior surgery
4. Stable tremor medication for at least 3 months prior inclusion
5. Written informed consent

Exclusion Criteria:

1. Major Depression with suicidal thoughts or suicidal thoughts in history
2. Dementia (Mattis Dementia Rating Score ≤ 130)
3. Acute psychosis
4. Patient incapability
5. Nursing care at home
6. Surgical contraindications
7. Medications that are likely to cause interactions in the opinion of the investigator
8. Known or persistent abuse of medication, drugs or alcohol
9. Persons who are in a relationship of dependence/employment with the sponsor or the investigator
10. Fertile women not using adequate contraceptive methods: female condoms, diaphragm or coil, each used in combination with spermicides; intra-uterine device; hormonal contraception in combination with a mechanical method of contraception;
11. Current or planned pregnancy, nursing period

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Tremor reduction defined by the difference in FTMTRS at 6 months after intervention to baseline | Baseline, 6 months after neurosurgery
  Tremor reduction defined by the difference in Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) at 6 months after intervention to baseline

SECONDARY OUTCOMES:
Effective tremor reduction at 12 months after intervention | Baseline, 12 months after neurosurgery
  Effective tremor reduction (an FTMTRS score reduction by 50% compared to baseline is regarded as "response") at 12 months after intervention
Tremor reduction measured by tremor analysis at baseline and 6 and 12 months after intervention | Baseline, 6 and 12 months after neurosurgery
  Tremor reduction will be measured by tremor analysis (an accelerometric examination); Unit: Hertz (Hz)
Tremor reduction measured by calculation of total power at baseline and 6 and 12 months after intervention | Baseline, 6 and 12 months after neurosurgery
  Tremor reduction will be assessed during Electromyography (EMG) by the calculation of total power; Unit: mg², with g=9,81 m/s²
Quality of Life: QUEST, SF-36 | Baseline, 6 and 12 months after neurosurgery
  Quality of Life assessed by Quality of Life Essential Tremor Questionnaire (QUEST) and Short Form (36) Health Survey
Size of VAT | Day 0 (Day of neurosurgery)
  Size of Volume of activated tissue (VAT)
Effective contact position with respect to DRT and AC-PC coordinates | Day 0 (Day of neurosurgery)
  Effective contact position of stimulation electrodes (with respect to the Dentato-rubro-thalamic bundle (DRT) and anterior commissure (AC) - posterior commissure (PC) line (ACPC) coordinates)
Duration of neurosurgery | Day 0 (Day of neurosurgery)
  Duration of neurosurgery (time points of mounting frame, start surgery, stop surgery (= dismounting frame)
Changes in BDI | Baseline, 6 and 12 months after neurosurgery
  Psychiatric assessment: changes in Beck's Depression Inventory (BDI)
Assessment of (Serious) Adverse Events related to intervention | Up to 12 months after neurosurgery

CONTACTS AND LOCATIONS:
Overall Officials: Volker A Coenen, MD, Principal Investigator — University Hospital Freiburg
Locations (1):
- University of Freiburg - Medical Center - Dept. of Stereotactic and Functional Neurosurgery, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Zappia M, Albanese A, Bruno E, Colosimo C, Filippini G, Martinelli P, Nicoletti A, Quattrocchi G, Abbruzzese G, Berardelli A, Allegra R, Aniello MS, Elia AE, Martino D, Murgia D, Picillo M, Squintani G. Treatment of essential tremor: a systematic review of evidence and recommendations from the Italian Movement Disorders Association. J Neurol. 2013 Mar;260(3):714-40. doi: 10.1007/s00415-012-6628-x. Epub 2012 Aug 11. PMID 22886006
- [Background] Koller W, Biary N, Cone S. Disability in essential tremor: effect of treatment. Neurology. 1986 Jul;36(7):1001-4. doi: 10.1212/wnl.36.7.1001. PMID 2940473
- [Background] Chopra A, Klassen BT, Stead M. Current clinical application of deep-brain stimulation for essential tremor. Neuropsychiatr Dis Treat. 2013;9:1859-65. doi: 10.2147/NDT.S32342. Epub 2013 Dec 2. PMID 24324335
- [Background] Benabid AL, Pollak P, Gao D, Hoffmann D, Limousin P, Gay E, Payen I, Benazzouz A. Chronic electrical stimulation of the ventralis intermedius nucleus of the thalamus as a treatment of movement disorders. J Neurosurg. 1996 Feb;84(2):203-14. doi: 10.3171/jns.1996.84.2.0203. PMID 8592222
- [Background] Deistung A, Schafer A, Schweser F, Biedermann U, Turner R, Reichenbach JR. Toward in vivo histology: a comparison of quantitative susceptibility mapping (QSM) with magnitude-, phase-, and R2*-imaging at ultra-high magnetic field strength. Neuroimage. 2013 Jan 15;65:299-314. doi: 10.1016/j.neuroimage.2012.09.055. Epub 2012 Oct 2. PMID 23036448
- [Background] Lemaire JJ, Sakka L, Ouchchane L, Caire F, Gabrillargues J, Bonny JM. Anatomy of the human thalamus based on spontaneous contrast and microscopic voxels in high-field magnetic resonance imaging. Neurosurgery. 2010 Mar;66(3 Suppl Operative):161-72. doi: 10.1227/01.NEU.0000365617.41061.A3. PMID 20173566
- [Background] Coenen VA, Allert N, Madler B. A role of diffusion tensor imaging fiber tracking in deep brain stimulation surgery: DBS of the dentato-rubro-thalamic tract (drt) for the treatment of therapy-refractory tremor. Acta Neurochir (Wien). 2011 Aug;153(8):1579-85; discussion 1585. doi: 10.1007/s00701-011-1036-z. Epub 2011 May 8. PMID 21553318
- [Background] Coenen VA, Allert N, Paus S, Kronenburger M, Urbach H, Madler B. Modulation of the cerebello-thalamo-cortical network in thalamic deep brain stimulation for tremor: a diffusion tensor imaging study. Neurosurgery. 2014 Dec;75(6):657-69; discussion 669-70. doi: 10.1227/NEU.0000000000000540. PMID 25161000
- [Background] Coenen VA, Madler B, Schiffbauer H, Urbach H, Allert N. Individual fiber anatomy of the subthalamic region revealed with diffusion tensor imaging: a concept to identify the deep brain stimulation target for tremor suppression. Neurosurgery. 2011 Apr;68(4):1069-75; discussion 1075-6. doi: 10.1227/NEU.0b013e31820a1a20. PMID 21242831
- [Background] Torres CV, Manzanares R, Sola RG. Integrating diffusion tensor imaging-based tractography into deep brain stimulation surgery: a review of the literature. Stereotact Funct Neurosurg. 2014;92(5):282-90. doi: 10.1159/000362937. Epub 2014 Sep 18. PMID 25248076
- [Background] Klein JC, Barbe MT, Seifried C, Baudrexel S, Runge M, Maarouf M, Gasser T, Hattingen E, Liebig T, Deichmann R, Timmermann L, Weise L, Hilker R. The tremor network targeted by successful VIM deep brain stimulation in humans. Neurology. 2012 Mar 13;78(11):787-95. doi: 10.1212/WNL.0b013e318249f702. Epub 2012 Feb 29. PMID 22377809
- [Derived] Sajonz BE, Amtage F, Reinacher PC, Jenkner C, Piroth T, Katzler J, Urbach H, Coenen VA. Deep Brain Stimulation for Tremor Tractographic Versus Traditional (DISTINCT): Study Protocol of a Randomized Controlled Feasibility Trial. JMIR Res Protoc. 2016 Dec 22;5(4):e244. doi: 10.2196/resprot.6885. PMID 28007690